CLINICAL TRIAL: NCT06472544
Title: Trauma-informed Intervention for Rheumatoid Arthritis on Blackfeet Nation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blackfeet Community College (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1674119
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Masking Description: As there is only one group which the intervention group there is no need for masking as to treatment type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Culturally Grounded Intervention (Experimental): One week of meetings to describe Blackfeet history, culture, traditions, and cerimonies. One additional week of visiting Blackfeet sacred sites.
  Interventions: Behavioral: Culturally Grounded Intervention

INTERVENTIONS:
Behavioral: Culturally Grounded Intervention — Education to increase awareness of Blackfeet culture and connectedness to Blackfeet community

SUMMARY:
The goal of this study is to determine whether an intervention grounded in Blackfeet culture improves systemic inflammation and symptoms of arthritis in Blackfeet People with rheumatoid arthritis. The intervention is designed to increase conectedness of Blackfeet people to Blackfeet culture and community. The intervention will consist of one week of meetings in which Blackfeet Elders talk about Blackfeet historical trauma, culture, traditions and cerimonies. The second week of the intervention consists of visiting Blackfeet sacred sites, guided by Blackfeet Elders. Participants will complete surveys to determine their conectedness to Blackfeet Culture, level of stress, Adverse Childhood Experiences Score (ACES) and arthritis symptoms. Participants will also be evaluated for clinical severity of arthritis and biomarkers of systemic inflammation. Participants will be evaluated pre- and post-intervention as well as 6 months post-intervention.

DETAILED DESCRIPTION:
The prevalence rate of rheumatoid arthritis (RA) in Blackfeet Nation members is among the highest in North America. With our current NARCH funding, we have found that cultural connectiveness in members of the Blackfeet Nation ameliorated the pro-inflammatory effects associated with high exposure to adverse childhood experiences (ACES). This raises the question of whether improving cultural connectedness might be an effective, trauma-informed approach to improve function, outcome, and/or a sense of well-being in individuals with rheumatic diseases such as RA. The plausibility of taking this approach is grounded on the high exposure rates to ACEs in individuals living on and near the Blackfeet Reservation and the strong association between ACEs and systemic inflammation. Thus, we will test the hypothesis that a trauma-informed intervention aimed to improve cultural connectiveness will improve subjective and objective features of RA in individuals living on or near the Blackfeet Nation Reservation. This research project will serve the overall goal of the NARCH grant by: (1) building on past NARCH research to better understand physical and mental health of the Blackfeet Nation; (2) building capacity for health research at BCC-CCM through engagement and training of BCC students, driving scholarly productivity of BCC faculty, and building new inter-institutional collaborations; and (3) generate compelling results to address health concerns for the Blackfeet Nation. We propose 2 aims that can be accomplished over the time frame of this application:

Specific Aim 1: We will test the effects of a 2-week intervention designed to connect individuals with RA more strongly to Blackfeet language, cultures, ceremonies, and land. This pilot intervention of limited size will consist of assessing the clinical symptoms of RA, ACES scores, and biomarkers of inflammation before and immediately after the culturally grounded intervention. This pilot will inform a second, more encompassing intervention in aim 2. Specific Aim 2: We will test the hypothesis that a 2-week intervention to improve cultural connectedness in individuals with RA living on or near the Blackfeet Nation result in objective changes to pro-inflammatory markers, including markers associated with disease activity in RA. We believe developing an intervention which could reduce systemic inflammation could not only ameliorate symptoms of RA but possibly other inflammation-mediated diseases as well.

ELIGIBILITY:
Inclusion Criteria: Diagnosis or self reporting of rheumatoid arthritis or use of rheumatoid arthritis medications.

Self reported Blackfeet heritage. -

Exclusion Criteria: Children under 18 years of age.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Rheumatoid Arthritis Disease Activity | Outcomes will be determined just before the intervention (day 1), just after intervention (day 14) and 6 months later.
  Arthritis activity will be determined bu clinical assessments and self-reported symptom severity.

SECONDARY OUTCOMES:
Systemic Inflammation | Systemic inflammation determined immediately before intervention (day 1), immediately after end of intervention 9Day 14), and 6 months after intervention.
  Systemic inflammation determined by assessing blood levels of inflammation biomarkers CRP, IL-6 and IL-17.

IPD SHARING:
Plan to Share IPD: No